CLINICAL TRIAL: NCT01356368
Title: A Pilot Study of Customizing First Line Chemotherapy in Advanced Non-Small Cell Lung Cancer Based on Molecular Markers
Brief Title: Customizing First Line Chemotherapy in Advanced Non-Small Cell Lung Cancer
Acronym: Customizing
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual rate
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC09/095
Record Dates: First submitted 2011-03-19; First posted 2011-05-19 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Cisplatin; Gemcitabine; Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cisplatin,Docetaxel,Gemzar, Premetrexed (Experimental): Patients will receive treatment for up to six cycles of the assigned regimen unless there is disease progression or unacceptable toxicities. After treatment, the patients will be seen every 2 months for the first year, then every 3 months for the second year and every 6 months afterwards.
  Interventions: Drug: Cisplatin, Gemzar, Docetaxel, Alimta

INTERVENTIONS:
Drug: Cisplatin, Gemzar, Docetaxel, Alimta — Patients will be assigned to treatment according to the molecular biological results which will analyze excision repair cross-complementing (ERCC1), ribonucleotide reductase subunit M1 (RRM1) and beta-tubulin genes in primary tumor cells which are present in tissues and peripheral blood.

SUMMARY:
The study aims at piloting the concept of customization of chemotherapy based on molecular markers in patients with stage IIIB (with pleural effusion) and IV with performance status ≤ 2 with pathologically proven non-small cell lung cancer (NSCLC). The study will not test or compare individual regimen but rather it will test the approach of customization concept as a whole.

The results of this pilot study will help in designing more definitive trials in our patient population.

DETAILED DESCRIPTION:
The treatment of advanced NSCLC cancer includes various chemotherapies with equivalent regimens that have reached a therapeutic plateau. The selection of these regimens is completely empirical and physician dependent. Potential predictors of specific agent efficacy exist in the form of tumor molecular markers that are a reflection of the individual's genetic make up. Thus our study aims at utilizing these markers to more efficiently select the regimen in order to maximize the benefit to the patients rather than using empiric approaches. Fortunately, each of our selected regimens contains active and well-studied agents in the treatment of lung cancer (Table 1). This pilot study will help us determine the benefit, and safety of this approach (not individual regimen). The study is not to compare individual regimens but it aims at testing the whole concept of customization of chemotherapy based on molecular markers to help us in the future at selecting regimens based on these markers and not empirically. The results then will be used to determine more definitive future studies.

Furthermore, circulating tumor cells in the blood represent the future distant metastases that result in disease progression to incurable stages. The circulating tumor cells have the ability to cross into vessels, travel in circulation, and exit the vessels into tissues where they have the capability to grow. Therefore, these cells may express different biological and molecular features from the stationary cells in the primary tumors. Therefore, exploiting these circulating tumor cells for augmenting treatment approaches is of vital importance and utility.

ELIGIBILITY:
Inclusion Criteria:

1. Microscopic diagnosis of NSCLC stages IIIB (with malignant pleural effusion) and IV
2. Having adequate tissue sample to perform the markers testing
3. Age ≥ 18 years
4. No prior chemotherapy treatment for lung cancer (Surgery and radiotherapy are acceptable)
5. No other concurrent cancer treatment
6. Performance status of 0- 2 per ECOG scale (Appendix II)
7. Adequate laboratory values as follows as follows:

   Absolute neutrophil count ≥ 1500/mm3 Platelet count ≥100, 000/ mm3 Total bilirubin ≤ 1.25X institutional upper normal level AST and ALT ≤ 3 X institutional upper normal level Serum creatinine ≤ 1.5 X institutional upper normal level
8. Presence of measurable disease

Exclusion Criteria:

1. Prior systemic treatment for lung cancer
2. History of hypersensitivity to drugs used
3. Diagnosis of other malignancy in the last 5 years excluding curatively treated non-melanoma skin cancer and in-situ cervical cancer
4. Medical illness that puts the patient at significant risk per investigator's discretion
5. Uncontrolled CNS disease. Patients with CNS metastatic disease treated with radiotherapy or surgery will be eligible if the CNS disease is stable 4 weeks after the treatment initiation without increase dose of steroids
6. Positive pregnancy test or refusal to use contraception during treatment. (Gynecology consultant for contraception)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Efficacy and Safety | 3 years
  1. Efficacy is measured by:
     * overall response rate (partial response and complete response) using RECIST Criteria
     * time to disease progression (TTP)
     * progression free survival (PFS)
     * overall survival (OS)
  2. To evaluate the Number of participants with Adverse Events and Serious Adverse Events.Safety will include 5 parameters to be collected for all patients who receive the study regimen which are:
     * Adverse Events
     * Laboratory Assessments
     * Vital Signs
     * Physical Examinations
     * ECG

SECONDARY OUTCOMES:
Tumor marker | 3 years
  1. The molecular characteristics of circulating tumor cells harvested from peripheral blood
  2. Correlation between the markers of circulating tumor cells and primary tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahman Jazieh, MD/MPH, Principal Investigator — King Abdul Aziz Medical City for National Guard
Locations (1):
- King Abdul Aziz Medical City for National Guard Health Affairs, Riyadh, Saudi Arabia